CLINICAL TRIAL: NCT01156272
Title: 3f 19mm IDE Study Rev D
Brief Title: Post Market ATS 3f® Aortic Bioprosthesis, Model 1000, Size 19mm
Status: Withdrawn | Type: Observational
Why Stopped: Study terminated prematurely.
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009
Record Dates: First submitted 2010-06-28; First posted 2010-07-02 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Heart Valve Diseases
Keywords: Isolated aortic valve replacement; heart valve
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Replacement aortic heart valve: ATS 3f® Aortic Bioprosthesis, Model 1000, Size 19mm
  Interventions: Device: ATS Medical 3f® Aortic Bioprosthesis, Model 1000 19mm

INTERVENTIONS:
Device: ATS Medical 3f® Aortic Bioprosthesis, Model 1000 19mm — Replacement aortic heart valve
  Other Names: Model 1000, 19mm

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the ATS 3f® Aortic Bioprosthesis, Model 1000 (Equine Pericardial Bioprothesis) size 19mm in a patient population undergoing isolated aortic valve replacement of his/her native aortic valve, or replacement of a failed prosthesis.

DETAILED DESCRIPTION:
A multi-center, post market, non-randomized trial, designed to obtain safety and efficacy data from patients implanted with the size 19mm Model 1000 heart valve. Each enrolled patient will be followed until one year post-implantation. Data will be collected both retrospectively and prospectively, on patients who were implanted from 1-Jan-2009 to 31-Dec-2009 with the 19mm Model 1000. The data collected will be pooled with the data currently collected, under the U.S. Food and Drug Administration (FDA) IDE Number G01284 for submission to the U.S. FDA.

ELIGIBILITY:
Inclusion Criteria:

* The patient required isolated aortic valve replacement with or without concomitant procedures such as coronary artery bypass or another valve reconstruction with an ATS 3f® Aortic Bioprosthesis Model 1000 (size 19mm) between the dates of 1-Jan-2009 and 31-Dec-2009. The three remaining heart valves must be of native tissue.
* The patient is geographically stable and willing to return to the implant center for any required follow-up visits.
* The patient has been adequately informed and consents to his/her participation in the clinical study, and of what will be required of him/her, in order to comply with the protocol.

Exclusion Criteria:

* The patient is twenty (20) or less than twenty years of age.
* The patient is an intravenous drug and/or alcohol abuser.
* The patient presented for implant with active endocarditis.
* The patient presented for implant with congenital bicuspid aortic anatomy.
* The patient had a previously implanted prosthetic valve that was not replaced by the study valve.
* The patient required mitral, tricuspid or pulmonic valve replacement.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were previously implanted with the ATS 3f Aortic Bioprosthesis Model 1000 (size 19mm) between the dates 1-Jan-2009 and 31-Dec-2009 and who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
New York Heart Association (NYHA) Functional Classification | <30 days / discharge, whichever comes last, 3-6 months, 11-14 months
  The NYHA classifications will be analyzed to demonstrate if implanting the of the study valve leads to an improvement in this clinical parameter for the patient.
Blood Data | <30 days / discharge, whichever comes last, 3-6 months, 11-14 months
  Blood data will be analyzed preoperative and postopertive to demonstrate if implanting of the study valve results in acceptable parameters for Serum Lactate Dehydrogenase (SLDH), Haptoglobin, Hematocrit and Reticulocyte parameters. Platelet and white blood cell count will also be analyzed.
Adverse/complication rates | <30 days / discharge, whichever comes last, 3-6 months, 11-14 months
  To demonstrate that the adverse/complication rates for the Model 1000 Bioprosthesis are less than two times the Objective Performance Criteria (OPCs) established by the FDA for severe complications.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Boulware, PhD, Study Director — Medtronic
Locations (1):
- McGill University Health Centre, Royal Victoria Hospital, Montreal, Quebec, Canada

REFERENCES:
- See also: Corporate Website — http://www.medtronic.com/